CLINICAL TRIAL: NCT00959647
Title: An Open-label, Multicenter Extension Study of GDC-0449 (Hedgehog Pathway Inhibitor) in Patients Treated With GDC-0449 in a Previous Genentech-sponsored Phase I or Phase II Cancer Study
Brief Title: A Study of Vismodegib (GDC-0449) in Patients Treated With Vismodegib in a Previous Genentech-sponsored Phase I or II Cancer Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHH4437g; GO01352 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-08-10; First posted 2009-08-14 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Ovarian Cancer; Basal Cell Carcinoma; Metastatic Colorectal Cancer
Keywords: Hedgehog pathway inhibitor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Basal Cell; Colorectal Neoplasms | interventions — HhAntag691; Folfox protocol; IFL protocol; Bevacizumab

ARMS (1):
- Vismodegib 150 mg (Experimental): Participants received 150 mg vismodegib orally once a day until disease progression, intolerable toxicity, or withdrawal from the study. If a participant had been receiving combination chemotherapy and/or biotherapy (FOLFOX, FOLFIRI, bevacizumab) in a parent study, the same combination chemotherapy and/or biotherapy as specified in the parent study could be continued in this study at the discretion of the investigator.
  Interventions: Drug: Vismodegib; Drug: FOLFOX; Drug: FOLFIRI; Drug: Bevacizumab

INTERVENTIONS:
Drug: Vismodegib — Vismodegib was supplied in capsules.
  Other Names: Erivedge; GDC-0449; RO5450815
Drug: FOLFOX — FOLFOX (folinic acid [FOL, leucovorin], fluorouracil [F, 5-FU], and oxaliplatin [OX]) was supplied as solutions for intravenous administration.
Drug: FOLFIRI — FOLFIRI (folinic acid [FOL, leucovorin], fluorouracil [F, 5-FU], and irinotecan [IRI]) was supplied as solutions for intravenous administration.
Drug: Bevacizumab — Bevacizumab was supplied as a solution for intravenous administration.
  Other Names: Avastin

SUMMARY:
This was a multicenter, open-label extension study. Patients who received vismodegib (GDC-0449) in a Genentech-sponsored study and who had completed the parent study or who continued to receive vismodegib at the time the parent study closed were eligible for continued treatment in this protocol.

ELIGIBILITY:
This study only enrolled participants who took part in previous studies of vismodegib conducted by Genentech.

Inclusion Criteria:

* Completed vismodegib treatment within 2-4 weeks in a Genentech-sponsored parent study or continued to receive vismodegib at the time the Genentech-sponsored parent study closed.
* Expectation by the investigator that the participant may continue to benefit from additional vismodegib treatment.

Exclusion Criteria:

* Intervening anti-tumor therapy not specified in the parent study (ie, non-protocol-specified chemotherapy, other targeted therapy, radiation therapy, or photodynamic therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josina Reddy, MD, PhD, Study Director — Genentech, Inc.
Locations (10):
- United States (10):
  - Scottsdale, Arizona
  - Oakland, California
  - Palm Springs, California
  - Stanford, California
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Las Vegas, Nevada
  - Cincinnati, Ohio
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vismodegib 150 mg
Started | 19
Completed | 0
Not Completed | 19
Not completed — Adverse Event | 2
Not completed — Progressive disease | 6
Not completed — Study terminated by sponsor | 4
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who had received at least 1 dose of study medication.
Arm/Group | Vismodegib 150 mg
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15

OUTCOME MEASURES:

1. Secondary Outcome: Incidence and Severity of All Adverse Events and Serious Adverse Events
Time Frame: 30 days following the last administration of study treatment
Reporting Status: Not Posted

2. Secondary Outcome: Incidence of Adverse Events Leading to GDC-0449 Discontinuation
Time Frame: 30 days following the last administration of study treatment
Reporting Status: Not Posted

3. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event
Time Frame: Baseline until 30 days following the last administration of study treatment
Population: Safety population: All participants who had received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Vismodegib 150 mg
Number analyzed (Participants) | 19
Percentage of participants | 89.5

4. Primary Outcome: Percentage of Participants Who Discontinued Treatment Due to an Adverse Event
Time Frame: Baseline until 30 days following the last administration of study treatment
Population: Safety population: All participants who had received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Vismodegib 150 mg
Number analyzed (Participants) | 19
Percentage of participants | 10.5

ADVERSE EVENTS:
Time Frame: From Baseline until 30 days following the last administration of study treatment.
Description: Safety population: All participants who had received at least 1 dose of study medication.
Arm/Group | Vismodegib 150 mg
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib 150 mg (N=19)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Tubo-ovarian abscess (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib 150 mg (N=19)
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Hernia (General disorders) | 1
Influenza like illness (General disorders) | 1
Local swelling (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Polyp (General disorders) | 1
Swelling (General disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 1
Weight decreased (Investigations) | 6
Hepatic enzyme increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Lactose intolerance (Metabolism and nutrition disorders) | 1
Dysgeusia (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Insomnia (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Anaemia macrocytic (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Purulent discharge (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Dry eye (Eye disorders) | 1
Eyelid cyst (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haematuria (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Urinary straining (Renal and urinary disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Seasonal allergy (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.